CLINICAL TRIAL: NCT02138097
Title: A Description of Oral and Non-insulin Injected Hypoglycemic Therapy Utilization Patterns Including Initiation, Switching, and Discontinuation
Brief Title: Oral and Non-insulin Injected Hypoglycemic Therapy Utilization Patterns
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218.161
Record Dates: First submitted 2014-05-13; First posted 2014-05-14 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (8):
- Glitazones
- Linagliptin
- Meglitinides
- Metformin
- Non-insulin injectables
- Saxagliptin
- Sitagliptin
- Sulfonylurea

SUMMARY:
This protocol is for a series of descriptive analyses conducted within a cohort of patients using linagliptin, other dipeptidyl peptidase-4 (DPP-4) inhibitors, and other oral and non-insulin injected hypoglycemic medications between May 2011 and July 2012.

Understanding 1) the existing utilization patterns for linagliptin, sitagliptin, saxagliptin, and other oral and non-insulin injected hypoglycemic agents and (2) the differences in utilization patterns between these agents will help with the design, analysis and interpretation of comparative effectiveness and safety studies of linagliptin, other DPP-4 inhibitors, and other agents.

The study will provide an overview of existing utilization patterns for linagliptin, other dipeptidyl peptidase-4 (DPP-4) inhibitors, other oral and non-insulin injected hypoglycemic agents, in order to detect potential selective prescribing patterns that might lead to channeling bias.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of type 2 diabetes mellitus
* a dispensing of an oral or non-insulin injected hypoglycemic medication between May 2011 and June 2012
* at least 6 months enrolment in the database preceding the date of the first dispensing

Exclusion criteria:

* age < 18
* missing or ambiguous age or sex information
* at least one diagnosis of type 1 diabetes mellitus or secondary diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM patients aged 18 years or older, initiating antidiabetic treatment after at least 6 months of continuous enrollment
Sampling Method: Non-Probability Sample
Enrollment: 615067 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1218.161.1 Boehringer Ingelheim Investigational Site, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Existing data cohort design using data from the United Healthcare and MarketScan databases from May 2011 through July 2012
Groups:
- United Healthcare: Patients using an oral and non-insulin injected glucose-lowering medication identified from the United Healthcare Research database
- MarketScan: Patients using an oral and non-insulin injected glucose-lowering medication identified from the MarketScan database.
Period: Overall Study
Arm/Group | United Healthcare | MarketScan
Started | 155345 | 459722
Completed | 155345 | 459722
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients included in the study
Groups:
- UHC: Glitazones: Patients in the United Healthcare cohort (UHC) using Glitazones as an oral and non-insulin injected glucose-lowering medication.
- UHC: Linagliptin: Patients in the United Healthcare cohort using Linagliptin as an oral and non-insulin injected glucose-lowering medication.
- UHC: Meglitinides: Patients in the United Healthcare cohort using Meglitinides as an oral and non-insulin injected glucose-lowering medication.
- UHC: Metformin: Patients in the United Healthcare cohort using Metformin as an oral and non-insulin injected glucose-lowering medication.
- UHC: Saxagliptin: Patients in the United Healthcare cohort using Saxagliptin as an oral and non-insulin injected glucose-lowering medication.
- UHC: Sitagliptin: Patients in the United Healthcare cohort using Sitagliptin as an oral and non-insulin injected glucose-lowering medication.
- UHC: Sulfonylurea: Patients in the United Healthcare cohort using Sulfonylurea as an oral and non-insulin injected glucose-lowering medication.
- UHC: Alpha-Glucosidase Inhibitors: Patients in the United Healthcare cohort using Alpha-Glucosidase Inhibitors (AGI) as an oral and non-insulin injected glucose-lowering medication.
- UHC: GLP-I RA: Patients in the United Healthcare cohort using glucagon-like peptide-1 (GLP-1) receptor agonists (RA) as an oral and non-insulin injected glucose-lowering medication.
- MS: Linagliptin: Patients in the MarketScan (MS) cohort using Linagliptin as an oral and non-insulin injected glucose-lowering medication.
- MS: Sitagliptin: Patients in the MarketScan (MS) cohort using Sitagliptin as an oral and non-insulin injected glucose-lowering medication.
- MS: Saxagliptin: Patients in the MarketScan (MS) cohort using Saxagliptin as an oral and non-insulin injected glucose-lowering medication.
- MS: Metformin: Patients in the MarketScan (MS) cohort using Metformin as an oral and non-insulin injected glucose-lowering medication.
- MS: Sulfonylurea: Patients in the MarketScan (MS) cohort using Sulfonylurea as an oral and non-insulin injected glucose-lowering medication.
- MS: Glitazones: Patients in the MarketScan (MS) cohort using Glitazones as an oral and non-insulin injected glucose-lowering medication.
- MS: Meglitinides: Patients in the MarketScan (MS) cohort using Meglitinides as an oral and non-insulin injected glucose-lowering medication.
- MS: Alpha-Glucosidase Inhibitors: Patients in the MarketScan (MS) cohort using Alpha-Glucosidase Inhibitors (AGI) as an oral and non-insulin injected glucose-lowering medication.
- MS: GLP-I RA: Patients in the MarketScan (MS) cohort using glucagon-like peptide-1 (GLP-1) receptor agonists (RA) as an oral and non-insulin injected glucose-lowering medication.
- Total: Total of all reporting groups
Arm/Group | UHC: Glitazones | UHC: Linagliptin | UHC: Meglitinides | UHC: Metformin | UHC: Saxagliptin | UHC: Sitagliptin | UHC: Sulfonylurea | UHC: Alpha-Glucosidase Inhibitors | UHC: GLP-I RA | MS: Linagliptin | MS: Sitagliptin | MS: Saxagliptin | MS: Metformin | MS: Sulfonylurea | MS: Glitazones | MS: Meglitinides | MS: Alpha-Glucosidase Inhibitors | MS: GLP-I RA | Total
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 495 | 10490 | 7708 | 58769 | 24550 | 205213 | 104422 | 22310 | 5412 | 1918 | 29420 | 615067
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.67 (9.99) | 55.90 (10.06) | 57.08 (10.46) | 52.57 (10.56) | 53.68 (9.66) | 54.40 (10.16) | 53.75 (10.40) | 55.93 (10.67) | 52.35 (9.54) | 58.72 (11.66) | 58.42 (11.98) | 56.84 (11.39) | 55.91 (12.08) | 57.94 (12.49) | 57.40 (11.66) | 62.50 (12.60) | 59.96 (12.00) | 54.28 (10.02) | 55.05 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2679 | 1175 | 505 | 32251 | 3400 | 7600 | 13631 | 201 | 5521 | 3368 | 26158 | 10838 | 97105 | 45668 | 9181 | 2526 | 909 | 16077 | 278793
  Male | 4524 | 1645 | 679 | 40443 | 4700 | 10891 | 20237 | 294 | 4969 | 4340 | 32611 | 13712 | 108108 | 58754 | 13129 | 2886 | 1009 | 13343 | 336274

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Initiators for United Healthcare Patients
Description: Number of patients initiating each individual agent divided by the number of patients initiating any oral or non-insulin injected hypoglycemic agent.
Time Frame: up to 12 months
Population: All subjects in the United Healthcare cohort
Measure: Number; unit: Percentage of participants
Groups:
- Glitazones: Patients using Glitazones as an oral and non-insulin injected glucose-lowering medication.
- Linagliptin: Patients using Linagliptin as an oral and non-insulin injected glucose-lowering medication.
- Meglitinides: Patients using Meglitinides as an oral and non-insulin injected glucose-lowering medication.
- Metformin: Patients using Metformin as an oral and non-insulin injected glucose-lowering medication.
- Saxagliptin: Patients using Saxagliptin as an oral and non-insulin injected glucose-lowering medication.
- Sitagliptin: Patients using Sitagliptin as an oral and non-insulin injected glucose-lowering medication.
- Sulfonylurea: Patients using Sulfonylurea as an oral and non-insulin injected glucose-lowering medication.
- Alpha-Glucosidase Inhibitors: Patients using Alpha-Glucosidase Inhibitors (AGI) as an oral and non-insulin injected glucose-lowering medication.
- GLP-I RA: Patients using glucagon-like peptide-1 (GLP-1) receptor agonists (RA) as an oral and non-insulin injected glucose-lowering medication.
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 495 | 10490
Percentage of participants
  Naive new users | 2.8 | 0.5 | 0.2 | 69.9 | 2.3 | 5.8 | 16.3 | 0.1 | 2.1
  Non-naive new users | 6.5 | 3.1 | 1.3 | 23.0 | 8.2 | 18.2 | 27.5 | 0.5 | 11.6
  Monotherapy | 2.4 | 1.2 | 0.4 | 67.4 | 2.5 | 6.0 | 15.9 | 0.2 | 4.1
  Dual Therapy | 3.8 | 1.3 | 0.3 | 41.8 | 6.3 | 13.6 | 28.5 | 0.1 | 4.3
  Other initiation other than mono- or dual therapy | 10.0 | 3.7 | 2.1 | 13.0 | 9.1 | 21.3 | 24.5 | 0.9 | 15.3

2. Primary Outcome: Proportion of Initiators for MarketScan Patients
Description: as for outcome 1
Time Frame: up to 12 months
Population: All subjects in MarketScan cohort
Measure: Number; unit: Percentage of participants
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 22310 | 7708 | 5412 | 205213 | 24550 | 58769 | 104422 | 1918 | 29420
Percentage of participants
  Naive new users | 3.0 | 0.4 | 0.4 | 69.1 | 2.1 | 5.9 | 17.2 | 0.1 | 1.6
  Non-naive new users | 6.5 | 2.8 | 1.9 | 23.2 | 8.1 | 18.8 | 27.5 | 0.7 | 10.6
  Monotherapy | 2.5 | 1.0 | 0.6 | 66.1 | 2.6 | 6.3 | 17.4 | 0.2 | 3.4
  Dual Therapy | 5.1 | 1.7 | 1.0 | 34.0 | 6.6 | 15.6 | 29.7 | 0.3 | 5.8
  Other initiation other than mono- or dual therapy | 9.6 | 3.0 | 2.7 | 16.9 | 9.0 | 21.8 | 21.4 | 1.1 | 14.5

3. Primary Outcome: Treatment Switching for United Healthcare Patients
Description: Number of patients with dispensing of a new non-insulin hypoglycemic agent without subsequent to the end of days' supply of the original agent plus 30 days
Time Frame: up to 12 months
Population: All subjects in United Healthcare cohort
Measure: Number; unit: participants/1000 participant years
Groups:
- Other DPP-4I: Patients using other dipeptidyl peptidase-4 inhibitors (DPP-4I) as an oral and non-insulin injected glucose-lowering medication.
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 25940 | 495 | 10490
participants/1000 participant years | 117.76 | 71.64 | 122.97 | 30.47 | 57.38 | 103.09 | 46.89 | 87.6 | 126.83 | 77.9

4. Primary Outcome: Treatment Switching for MarketScan Patients
Description: as for outcome 3
Time Frame: up to 12 months
Population: All subjects in MarketScan cohort
Measure: Number; unit: participants/1000 participant years
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 22310 | 7708 | 5412 | 205213 | 24550 | 58769 | 104422 | 81760 | 1918 | 29420
participants/1000 participant years | 110.35 | 72.48 | 96.88 | 27.81 | 60.31 | 52.25 | 40.87 | 54.33 | 102.9 | 67.1

5. Primary Outcome: Treatment Augmentation for United Healthcare Patients
Description: Number of patients dispensing of a new non-insulin hypoglycemic agent while continuing to fill prescriptions for the initial therapy
Time Frame: up to 12 months
Population: All patients in United Healthcare cohort
Measure: Number; unit: participants/1000 participant years
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 25940 | 495 | 10490
participants/1000 participant years | 308.04 | 274.68 | 331.17 | 204.43 | 269.02 | 340.69 | 252.08 | 317.89 | 330.95 | 199.60

6. Primary Outcome: Treatment Augmentation for MarketScan Patients
Description: as for outcome 5
Time Frame: up to 12 months
Population: All patients in MarketScan cohort
Measure: Number; unit: participants/1000 participant years
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 22310 | 7708 | 5412 | 205213 | 24550 | 58769 | 104422 | 81760 | 1918 | 29420
participants/1000 participant years | 310.93 | 309.36 | 269.53 | 201.04 | 275.57 | 237.31 | 226.11 | 248.28 | 287.85 | 184.84

7. Primary Outcome: Subsequent Insulin Initiation for United Healthcare Patients
Description: Number of patients filling an insulin prescription subsequently to initiation of the original non-insulin agent without having filled one in the past 6 months
Time Frame: up to 12 months
Population: All patients in United Healthcare cohort
Measure: Number; unit: participants/1000 participant years
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 25940 | 495 | 10490
participants/1000 participant years | 112.61 | 101.17 | 162.97 | 56.49 | 97.37 | 103.26 | 92.02 | 101.44 | 142.42 | 135.58

8. Primary Outcome: Subsequent Insulin Initiation for MarketScan Patients
Description: as for outcome 7
Time Frame: up to 12 months
Population: All patients in MarketScan cohort
Measure: Number; unit: participants/1000 participant years
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 22310 | 7708 | 5412 | 205213 | 24550 | 58769 | 104422 | 81760 | 1918 | 29420
participants/1000 participant years | 109.1 | 111.02 | 168.83 | 57.99 | 105.7 | 103.65 | 89.57 | 103.85 | 191.54 | 136.56

9. Secondary Outcome: Treatment Discontinuation for United Healthcare Patients
Description: Number of patients with a treatment gap of >=6 months (i.e., no dispensing of non-insulin hypoglycemic agents within 6 months after the end of days supplied)
Time Frame: up to 12 months
Population: All subjects in United Healthcare cohort
Measure: Number; unit: participants/1000 participant years
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 25940 | 495 | 10490
participants/1000 participant years | 523.32 | 287.61 | 466.55 | 293.23 | 267.60 | 267.75 | 288.55 | 266.83 | 479.31 | 337.30

10. Secondary Outcome: Treatment Discontinuation for Marketscan Patients
Description: as for outcome 9
Time Frame: up to 12 months
Population: All subjects in Marketscan cohort
Measure: Number; unit: participants/1000 participant years
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 22310 | 7708 | 5412 | 205213 | 24550 | 58769 | 104422 | 81760 | 1918 | 29420
participants/1000 participant years | 522.1 | 284.67 | 463.13 | 285.58 | 261.2 | 262.24 | 285.75 | 261.06 | 504.83 | 333.9

11. Secondary Outcome: Proportion of Days Covered for United Healthcare Patients
Description: Number of days supply dispensed divided by number of days followed
Time Frame: up to 12 months
Population: All patients in United Healthcare cohort
Measure: Mean (Standard Deviation); unit: days covered
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 25940 | 495 | 10490
days covered | 68.79 (19.68) | 77.54 (18.91) | 64.04 (19.94) | 70.37 (20.31) | 75.81 (19.30) | 73.09 (19.30) | 72.46 (20.58) | 74.03 (19.32) | 67.48 (19.62) | 68.34 (19.66)

12. Secondary Outcome: Proportion of Days Covered for MarketScan Patients
Description: Number of days supply dispensed divided by number of days followed
Time Frame: up to 12 months
Population: All patients in MarketScan cohort
Measure: Mean (Standard Deviation); unit: days covered
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 22310 | 7708 | 5412 | 205213 | 24550 | 58769 | 104422 | 81760 | 1918 | 29420
days covered | 72.04 (19.82) | 78.62 (19.15) | 69.58 (20.56) | 74.40 (20.20) | 78.13 (19.34) | 77.80 (19.78) | 76.09 (20.28) | 78.00 (19.61) | 69.82 (20.38) | 71.30 (20.23)

13. Secondary Outcome: Persistence at 3 Months for United Healthcare Patients
Description: Fraction of non-insulin hypoglycemic initiators with continued dispensing. Patients will be classified as persistent if they possess medication at 3 months. Grace period of 30 days will be allowed.
Time Frame: 3 months
Population: All patients in United Healthcare cohort
Measure: Number; unit: Percentage of participants
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 25940 | 495 | 10490
Percentage of participants | 68.90 | 82.84 | 59.12 | 70.63 | 81.40 | 77.27 | 73.2 | 78.79 | 65.86 | 68.98

14. Secondary Outcome: Persistence at 6 Months for United Healthcare Patients
Description: Fraction of non-insulin hypoglycemic initiators with continued dispensing. Patients will be classified as persistent if they possess medication at 6 months. Grace period of 30 days will be allowed.
Time Frame: 6 months
Population: All patients in United Healthcare cohort
Measure: Number; unit: Percentage of participants
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 25940 | 495 | 10490
Percentage of participants | 42.02 | 64.65 | 34.29 | 48.38 | 62.90 | 55.41 | 51.71 | 57.95 | 39.80 | 47.25

15. Secondary Outcome: Persistence at 12 Months for United Healthcare Patients
Description: Fraction of non-insulin hypoglycemic initiators with continued dispensing. Patients will be classified as persistent if they possess medication at 12 months. Grace period of 30 days will be allowed.
Time Frame: 12 months
Population: All patients in United Healthcare cohort
Measure: Number; unit: Percentage of participants
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 7203 | 2820 | 1184 | 72694 | 8100 | 18491 | 33868 | 25940 | 495 | 10490
Percentage of participants | 28.35 | 51.45 | 22.64 | 35.45 | 49.75 | 36.84 | 38.58 | 40.95 | 25.05 | 33.58

16. Secondary Outcome: Persistence at 3 Months for MarketScan Patients
Description: as for outcome 13
Time Frame: 3 months
Population: All patients in MarketScan cohort
Measure: Number; unit: Percentage of participants
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 22310 | 7708 | 5412 | 205213 | 24550 | 58769 | 104422 | 81760 | 1918 | 29420
Percentage of participants | 73.47 | 83.39 | 68.90 | 76.89 | 82.82 | 81.58 | 78.72 | 82.12 | 69.08 | 73.05

17. Secondary Outcome: Persistence at 6 Months for MarketScan Patients
Description: as for outcome 14
Time Frame: 6 months
Population: All patients in MarketScan cohort
Measure: Number; unit: Percentage of participants
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 22310 | 7708 | 5412 | 205213 | 24550 | 58769 | 104422 | 81760 | 1918 | 29420
Percentage of participants | 42.70 | 62.91 | 39.32 | 51.37 | 63.07 | 59.54 | 53.87 | 60.80 | 39.62 | 48.40

18. Secondary Outcome: Persistence at 12 Months for MarketScan Patients
Description: as for outcome 15
Time Frame: 12 months
Population: All patients in MarketScan cohort
Measure: Number; unit: Percentage of participants
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Number analyzed (Participants) | 22310 | 7708 | 5412 | 205213 | 24550 | 58769 | 104422 | 81760 | 1918 | 29420
Percentage of participants | 29.04 | 50.30 | 27.18 | 39.32 | 50.15 | 46.83 | 41.60 | 47.95 | 27.27 | 35.81

ADVERSE EVENTS:
Description: Serious and other (non-serious) adverse events were not of interest in this study and therefore were not collected or assessed as part of the study, in addition individual patient data is not available therefore adverse event data is not presented.
Arm/Group | Glitazones | Linagliptin | Meglitinides | Metformin | Saxagliptin | Sitagliptin | Sulfonylurea | Other DPP-4I | Alpha-Glucosidase Inhibitors | GLP-I RA
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.